CLINICAL TRIAL: NCT01545557
Title: Pan Facial Volume Restoration With a New Hyaluronic Acid Dermal Filler
Brief Title: Pan Facial Volume Restoration
Acronym: EVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.CIP.29090
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Volume Loss (Soft Tissue Ptosis or Atrophy )
Keywords: Volume loss
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronic acid dermal filler (Experimental): One Emervel Volume injection at baseline and touch up injections 3 weeks after if needed
  Interventions: Device: Hyaluronic acid dermal filler gel

INTERVENTIONS:
Device: Hyaluronic acid dermal filler gel — 1 Emervel Volume injection per indication and 1 touch-up injection if necessary
  Other Names: Study filler is Emervel Volume Lidocaine.

SUMMARY:
The aim of this study is to assess performance and tolerance as well as investigator and subject satisfaction further to pan-facial volume restoration with a new cross-linked hyaluronic acid dermal filler containing lidocaine 0.3%.

DETAILED DESCRIPTION:
Clinical hypothesis: The global approach of the subject pan-facial dermal volume depletion and face soft-tissue contour defects correction using specific dermal filler for all indications to be injected will satisfy both subjects and investigators.

This device will be used for full face correction of volume loss: chin, temporal areas, jawline, cheek, cheekbones, deep to very deep nasolabial folds (only if cheekbones are injected concomitantly).

Study duration will be up to 19 months. Injections will be performed at baseline. If necessary, investigator will perform touch-up injections at the following visit (3 weeks after baseline injection).

ELIGIBILITY:
Inclusion Criteria:

* Subjects seeking treatment for correction of volume loss.
* Subjects presenting a score of at least 2 (visible depression or descent) for whole face on the volume loss scale and at least 2 indications affected by volume loss among the following: chin temporal areas, jawlines, cheeks, cheekbones, deep to very deep nasolabial folds (severity score 4 at least on Lemperle rating scale) if cheekbones are injected.

Exclusion Criteria:

* Subjects at risk in term of precautions, warnings and contraindication referred in the package insert of the study device,
* Subjects who underwent previous injection of permanent filler in the injected area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2014-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist, Study Director — Galderma R&D
Locations (3):
- Brazil (3):
  - Galderma Investigational Center, Botucatu
  - Galderma Investigational Center, Rio de Janeiro
  - Galderma Investigational Center, Saö Paulo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty subjects were recruited across 4 sites in Brazil (15 subjects per site) between February 2012 and October 2013.
Groups:
- Hyaluronic Acid: Hyaluronic acid dermal filler gel: 1 injection per indication and 1 touch-up injection if necessary
Period: Overall Study
Arm/Group | Hyaluronic Acid
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 6
  Race: White | 53
  Race: Hispanic | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Volume Loss Assessment
Description: Overall loss of volume on full face was graded on a volume loss scale (VLS) of 0 to 3 by the investigator as follow: 0= normal, 1= evidence of early soft tissue ptosis or atrophy slightly visible, 2=visible depression or descent, 3= severe depression or atrophy. Last injections were given either at baseline or touch-up injections (if needed) on previously injected areas at 3 Weeks after baseline.
Time Frame: Baseline and 18 Months after last injection
Population: ITT population included all participants who were injected.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Volume loss18 Months After Injection: Full face volume loss 18 months after last injections for all subjects having received Hyaluronic Acid injections
Arm/Group | Volume loss18 Months After Injection
Number analyzed (Participants) | 60
Score on a scale | -0.8 (0.7)

2. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied at 3 Weeks After Last Injection
Description: Participants satisfaction with the overall, full face aesthetic results were assessed by use of participants global satisfaction questionnaire. Participants rated their satisfaction by answering question ; Rate overall, full face aesthetic outcome using the following options: not satisfied, somewhat satisfied, satisfied or very satisfied. Percentage of participants satisfied and very satisfied with the full face aesthetic outcome at 3 weeks after last injection were reported.
Time Frame: At 3 Weeks after last injection
Population: ITT population included all participants who were injected. Here, 'overall number of participants analyzed' signifies participants who completed a questionnaire about their satisfaction with the overall, full face aesthetic outcome.
Measure: Number; unit: Percentage of participants
Groups:
- Full Face Overall Aesthetic Outcome: All participants satisfied to very satisfied with overall full face aesthetic outcome
Arm/Group | Full Face Overall Aesthetic Outcome
Number analyzed (Participants) | 59
Percentage of participants
  Satisfied | 32.2
  Very satisfied | 67.8

3. Secondary Outcome: Percentage of Investigators Satisfied With the Use of Study Hyaluronic Acid Dermal Filler
Description: The study investigators (injectors) were requested to complete a questionnaire about their satisfaction with the use of study hyaluronic acid dermal filler (Emervel® Volume Lidocaine). The percentage of investigators who agreed to use Emervel® Volume Lidocaine again were reported in this outcome measure.
Time Frame: Baseline up to 18 Months after last injection
Population: Here overall number of participants analyzed refers to the study investigators who completed a questionnaire about their satisfaction with the use of study hyaluronic acid dermal filler.
Measure: Number; unit: percentage of participants
Groups:
- The Study Investigators (Injectors): The study investigators (injectors) who injected study product to the participants included in the study.
Arm/Group | The Study Investigators (Injectors)
Number analyzed (Participants) | 7
percentage of participants | 100

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 18 Months after last injection
Population: The safety population was defined as all participants who were injected with the study product.
Measure: Count of Participants; unit: Participants
Groups:
- Hyaluronic Acid: All injected participants.
Arm/Group | Hyaluronic Acid
Number analyzed (Participants) | 60
Participants | 9

5. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied at 18 Months After Last Injection
Description: Participants satisfaction with the overall, full face aesthetic results were assessed by use of participants global satisfaction questionnaire. Participants rated their satisfaction by answering question; rate overall, full face aesthetic outcome using the following options : not satisfied, somewhat satisfied, satisfied or very satisfied. Percentage of participants satisfied and very satisfied with the full-face aesthetic outcome at 18 Months after last injection were reported.
Time Frame: At 18 Months after last injection
Population: All injected subjects satisfied to very satisfied
Measure: Number; unit: percentage of participants
Groups:
- Full Face Overall Aesthetic Outcome: Percent of subjects satisfied to very satisfied with overall full face aesthetic outcome
Arm/Group | Full Face Overall Aesthetic Outcome
Number analyzed (Participants) | 60
percentage of participants
  Satisfied | 25
  Very satisfied | 70

ADVERSE EVENTS:
Time Frame: From Baseline up to 18 Months after last injection
Arm/Group | Hyaluronic Acid
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 2/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid (N=60)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) — unrelated to study product or injection procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of Institution and Investigator/Researcher to publish or disclose in any way Information requires Sponsor's prior written approval. Investigator/Researcher shall provide his draft of such publication to Sponsor for review and approval at least two months prior to the date of intended publication. Sponsor hereby agrees he shall endeavour to preserve accuracy of results in authorized publications and negative as well as positive results shall be published or made publicly available.